CLINICAL TRIAL: NCT01046526
Title: fMRI Study of Nicotinic Effect on Neurophysiology of Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905398; 05-DA-N398
Record Dates: First submitted 2010-01-09; First posted 2010-01-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-05-03

CONDITIONS: Schizophrenia; Psychopathology; Nicotine Dependence
Keywords: Psychopathology; Nicotine Patch; Eye Tracking; Attention; Schizophrenic Participants
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Individuals who have schizophrenia are significantly more likely to smoke than the general population, which leads to increased smoking-related illnesses and high rates of nicotine dependence. Research suggests that high rates of smoking and nicotine addiction in people with schizophrenia are related to the fact that nicotine temporally improves performance in several cognitive tasks, including sensory gating, long-term memory, and visual tracking-all of which are affected by schizophrenia.
* Smoking among schizophrenia patients may be a form of self-medication, since nicotine may temporarily treat and improve cognitive deficits caused by schizophrenia. Researchers are interested in studying the effects of nicotine on the brain activity of individuals with schizophrenia to better understand how nicotine affects the brain regions connected to memory, visual tracking, and attention.

Objectives:

* To identify specific brain regions involved in the anticipatory learning deficits found in schizophrenia patients who smoke.
* To determine whether and how nicotine enhances performance in these regions.

Eligibility:

- Smokers (at least 10 cigarettes per day) between 18 and 50 years of age who either are healthy volunteers or have been diagnosed with schizophrenia/schizoaffective disorder.

Design:

* Participants will be asked to avoid consuming alcohol and restrict consuming caffeinated beverages for 24 hours before the study days. Participants will provide urine and breath samples at the start of the study to be tested for chemicals that may interfere with the study.
* The study will require two to four visits, with two fMRI sessions and other visits for a clinical interview or training.

Participants will have a training session with a possible mock MRI scan to learn how to do tasks that track eye movement and measure ability to pay attention.

* During the fMRI scanning sessions, participants will receive either a nicotine patch or a placebo patch without nicotine. After the patch is in place, participants will perform tasks while receiving MRI scans. The scans will take up to 2 hours.
* Participants will provide blood samples after finishing the MRI sessions.

DETAILED DESCRIPTION:
The prevalence rate of smoking among schizophrenia patients is as high as 88 percent. This is associated with a 2-fold increase in deaths due to smoking related diseases-compounded by high rates of nicotine dependence and low abstinence rates following cessation programs. Converging lines of evidence suggest that high rates of smoking and nicotine addiction among schizophrenic patients is influenced by the presence of disease-related abnormalities in brain function. Genetic and post mortem studies show that patients exhibit abnormalities in neuronal nicotinic receptors, which are involved in a number of cognitive functions. Pharmacological studies show that nicotine temporally improves performance in several cognitive tasks including sensory gating, long-term memory, and visual tracking. These data support a growing consensus that smoking among schizophrenic patients is a form of self-medication, and suggest that the success of targeted smoking cessation programs will depend, in part, on finding alternative means of treating the underlying cognitive deficits. One of the most reproducible neurocognitive and biological changes in schizophrenia is abnormal visual tracking, or smooth pursuit eye movements. Preliminary data show that previously reported deficits in visual tracking are related to anticipatory learning deficits and that nicotine enhances performance in patients by temporarily treating this learning deficit. A better understanding of these processes may lead to better behavioral and/or pharmacological therapeutic interventions for excessive nicotine abuse and recidivism in this clinically vulnerable population. In order to identify brain regions underlying this learning deficit we propose to compare brain activations in 30 healthy controls and 30 patients with schizophrenia during anticipation of target motion using functional magnetic resonance imaging (fMRI). In order to identify the brain regions involved in nicotine-induced enhancement of anticipatory learning we will compare activation in patients under conditions of unexpected and anticipated target motion following administration of nicotine and placebo.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects (schizophrenia patients and healthy control smokers) must be between the ages of 18-50 and in good health based on history and physical exams. Age restrictions are based on age-related declines (usually occurring after age 55-58) in eye tracking performance. Schizophrenia patients are persons with a DSM-IV Axis-I diagnosis for schizophrenia, based on a best-estimate diagnosis by the Structured Clinical Interview for DSM-IV (SCID) supplemented by family informants and medical records, done at the MPRC. Those in nicotine protocols must demonstrate that they are experienced users based upon exhaled CO and must smoke a minimum of 10 cigarettes/day with duration of use of at least 1 year. Subjects may be users of alcohol and/or marijuana but may not meet criteria for dependence on either and may not have used either for at least 24 hours prior to scanning.

EXCLUSION CRITERIA:

Subjects will be excluded if they are unable to undergo MRI scanning due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or claustrophobia. Subjects will also be excluded if they have 1) any major medical illnesses to include, but not limited to, uncontrolled high blood pressure or high blood sugar, cardiovascular disease, asthma, peripheral vascular diseases, coagulopathies, history of superficial or deep vein thrombosis, HIV, or other infectious diseases (e.g. Hepatitis B), 2) mood or anxiety disorders, or substance-induced psychiatric disorders, 3) neurological illnesses to include, but not limited to, seizure disorders, multiple sclerosis, movement disorders, or history of head trauma, CVA, CNS tumor, and other conditions that cause neurocognitive sequelae, 4) significant alcohol or other drug use, other than nicotine dependence, 5) if their T1 weighted images reveal gross structural abnormalities and/or, 6)have a history of syncope. Urine pregnancy tests will be performed on all female volunteers of child-bearing age before each experimental session. Subjects who are positive for any drug other than nicotine or marijuana will be excluded. Subjects in nicotine protocols may not be actively seeking or engaged in smoking cessation treatment. If a subject requires change of antipsychotic medications because of exacerbation of psychotic symptoms, the subject will be considered clinically unstable and his/her participation will be discontinued. Patients with Axis-I mood disorders or substance-induced psychiatric disorders are excluded. We also exclude patients with significant alcohol or other illicit drug use, other than nicotine dependence. This is operationally defined as no SCID/DSM-IV Axis-I substance dependence in the past 6 months, and no current substance abuse. Exceptions are occasional use of marijuana.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-02-08; Study Completion 2012-05-03

CONTACTS AND LOCATIONS:
Overall Officials: George R Uhl, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Adam JJ, Backes W, Rijcken J, Hofman P, Kuipers H, Jolles J. Rapid visuomotor preparation in the human brain: a functional MRI study. Brain Res Cogn Brain Res. 2003 Mar;16(1):1-10. doi: 10.1016/s0926-6410(02)00204-5. PMID 12589883
- [Background] Adler LE, Hoffer LD, Wiser A, Freedman R. Normalization of auditory physiology by cigarette smoking in schizophrenic patients. Am J Psychiatry. 1993 Dec;150(12):1856-61. doi: 10.1176/ajp.150.12.1856. PMID 8238642
- [Background] Avila MT, Hong E, Thaker GK. Current progress in schizophrenia research. Eye movement abnormalities in schizophrenia: what is the nature of the deficit? J Nerv Ment Dis. 2002 Jul;190(7):479-80. doi: 10.1097/01.NMD.0000022450.48639.D3. No abstract available. PMID 12142851